CLINICAL TRIAL: NCT00579592
Title: A Pilot Study of Campath-1H Induction Therapy Combined With Rituximab®, Myfortic™ and a Short Course of Calcineurin Inhibitor Therapy to Allow for a Long Term Calcineurin Inhibitor Free Regimen After Renal Transplantation
Brief Title: Campath, Rituximab, and Myfortic With Short-Course Calcineurin Inhibitor Therapy in Renal Transplanation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Higher than expected rate of acute rejection
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2005-0454
Record Dates: First submitted 2007-12-17; First posted 2007-12-24 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Acute Rejection; Renal Transplantation
MeSH Terms: interventions — Alemtuzumab; Rituximab; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Campath, Rituximab, Myfortic, and 10-20 days of cyclosporine
  Interventions: Drug: Campath-1H, rituximab, myfortic

INTERVENTIONS:
Drug: Campath-1H, rituximab, myfortic — Campath-1H 30mg IV x 2 doses, rituximab 375mg/m2 IV x 1 dose, myfortic 720mg bid, cyclosporine po bid (target trough 200ng/ml) x 10-20 days

SUMMARY:
The hypothesis of this study is that lymphocyte depletion by Campath-1H and rituximab will obviate the need for long-term calcineurin inhibitors in renal transplantation. Most successful strategies to date have relied on the use of either tacrolimus or cyclosporine for an indefinite period of time. However, the advantage of a long term, calcineurin inhibitor free regimen may include improved renal allograft function, a lower incidence of hypertension, diabetes, and less drug related side effects. This is a non-randomized open-label pilot trial in 30 adult renal transplant patients. Subjects will receive 2 doses of Campath-1H (30mg given on Day 0 and Day 1) and a single dose of Rituximab (375mg/m2) on Day 0, given intra-operative. Subjects will take maintenance doses of prednisone and enteric coated mycophenolate sodium (Myfortic™). Subject will also be given cyclosporine (Neoral®) therapy for approximately 2 weeks (10-20 days).

ELIGIBILITY:
Inclusion Criteria:

* Recipient of cadaver or non HLA identical living donor transplantation (tx), Re-tx recipient (second tx) allowed, but no organ other than a kidney (ie no prev k/p)
* Females of CBP must have neg preg test at the time of study enrollment (SOC) & agree to practice birth control for duration of the study, or for 6 weeks after the last dose of Myfortic

Exclusion Criteria:

* Subjects who are pregnant or nursing.
* Current malignancy or a malignancy in the past 5 years, except for excised skin CA (BCC or SC)
* Multi-organ tx, ABO incompatible and + CM
* Subjects with a current PRA >50% within the past 30 days pre tx
* Subjects with active current infection requiring continued use of antibiotics, or the presence of chronic active hepatitis B (surface antigen +) or +HCV.
* Exclude for subjects who have received an investigational drug within 4 weeks of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-04; Primary Completion 2007-03 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
renal function | 2 years

SECONDARY OUTCOMES:
hypertension | 2 years
drug side effects | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hans Sollinger, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States